CLINICAL TRIAL: NCT03032874
Title: Colorectal Cancer Control in Low Resource Countries: Results From a Prospective Cohort Study of Patients at High-risk for Colorectal Cancer
Brief Title: Community Based Screening for Colorectal Cancer in an Underserved High Risk Population in Nigeria
Status: Completed | Type: Observational
Sponsor: Obafemi Awolowo University Teaching Hospital (Other)
Collaborators: Memorial Sloan Kettering Cancer Center, New York, USA (Unknown); University College Hospital, Nigeria (Unknown); University of Ilorin Teaching Hospital (Other)
Responsible Party: Principal Investigator, Olusegun Alatise, Consultant Surgeon/Senior Lecturer, Obafemi Awolowo University Teaching Hospital
Other Study IDs: ERC/2013/02/07
Record Dates: First submitted 2017-01-25; First posted 2017-01-26 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Polyps; Colonoscopy; Rectal bleeding; Nigeria
MeSH Terms: conditions — Colorectal Neoplasms; Polyps; Gastrointestinal Hemorrhage | interventions — Colonoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Colonic polyps and colorectal cancer specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Training set: All the patients with rectal bleeding who had colonoscopy performed at Obafemi Awolowo University Teaching Hospitals Complex
  Interventions: Procedure: Colonoscopy
- Validation set: All the patients with rectal bleeding who had colonoscopy performed at University College Hospital, Ibadan and University of Ilorin Teaching Hospital
  Interventions: Procedure: Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy — They all had screening colonoscopy

SUMMARY:
Patient age 45 year old and above who presented with rectal bleeding at three tertiary hospitals in South West Nigeria were invited for colonoscopy. The clinical information of the patients and the colonoscopy data were analyzed

DETAILED DESCRIPTION:
Patient age 45 year old and above who presented with rectal bleeding at Obafemi Awolowo University Teaching Hospitals Complex, Ile Ife, Nigeria, University College Hospital, Ibadan, Nigeria, and University of Ilorin Teaching Hospital, Ilorin Nigeria were invited for colonoscopy. Categorical variables were compared using χ2-test or Fisher's exact test while the Kruskal-Wallis test was used for quantitative variables. Multivariate analysis was performed using logistic regression model. All statistical tests were two-sided and p-values below 0.05 were considered statistically significant. Statistical analysis was carried out using SAS 9.4 and R 3.3.1.

ELIGIBILITY:
Inclusion Criteria:

* must be 45-years of age or older
* has rectal bleeding lasting at least one week
* has had a complete colonoscopy performed

Exclusion Criteria:

* Individuals with a personal history of inflammatory bowel disease, colorectal polyps, colorectal adenoma or CRC
* Individuals with a family history of familial adenomatous polyposis syndromes or other hereditary polyposis syndromes, hereditary nonpolyposis colorectal cancer
* Individuals with severe comorbidities that were contraindication to colonoscopy
* Individuals who had a previous history of colectomy

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Nigerians with rectal bleeding
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2016-07-30 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
To determine colonoscopy polyp and cancer detection rate | 2 years
  The hypothesis for this study was that colonoscopy surveillance of a high-risk cohort of patients with rectal bleeding would demonstrate that 10-20% of these patients have pre-malignant colorectal polyps(adenomas) or cancers.

SECONDARY OUTCOMES:
To detect colorectal cancer early using symptoms based assessment | 2 years
  The long-term impact of identifying at risk patients and patients with early stage cancers may be a reduction in mortality from colorectal cancer in low- and middle- income countries

CONTACTS AND LOCATIONS:
Locations (1):
- Endoscopy Unit, Obafemi Awolowo University Teaching Hospitals, Ile-Ife, Osun State, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided
Each request will be review on their merit by the team and approval of the Ethic and Research Committee that approve the study

REFERENCES:
- [Derived] Alatise OI, Ayandipo OO, Adeyeye A, Seier K, Komolafe AO, Bojuwoye MO, Afuwape OO, Zauber A, Omisore A, Olatoke S, Akere A, Famurewa O, Gonen M, Irabor DO, Kingham TP. A symptom-based model to predict colorectal cancer in low-resource countries: Results from a prospective study of patients at high risk for colorectal cancer. Cancer. 2018 Jul 1;124(13):2766-2773. doi: 10.1002/cncr.31399. Epub 2018 Apr 12. PMID 29645077